CLINICAL TRIAL: NCT01176305
Title: Venous Thromboembolism in Pregnant and Puerperal Women in Denmark 1995-2005
Status: Completed | Type: Observational
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Thomas Bergholt, Hillerod Hospital, Gynecolocical-Obstetrical department
Other Study IDs: RAV1
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2009-10

CONDITIONS: Venous Thromboembolism
Keywords: Thromboembolic event
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Danish Women 15 to 49 years old.: Free of previous VTE and current use of oral contraceptives.

SUMMARY:
The purpose of this study is to describe the incidence of thromboembolic events in relation to pregnancy and when in pregnancy and the puerperal period.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) still causes maternal death in the western world. The purpose of this study is to estimate the relative and absolute risk of VTE at different gestational ages in pregnant women compared to non-pregnant women.

All Danish Women 15 to 49 years old in the period January 1995 through December 2005, free of previous VTE and current use of oral contraceptives are included.Non-pregnant women are controls.

ELIGIBILITY:
Inclusion Criteria:

* Danish woman at 15 to 49 years old in the period January 1995 through December 2005.
* Free of previous VTE and current use of oral contraceptives.

Exclusion Criteria:

* Previous VTE or current use of oral contraceptives.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Danish Women 15 to 49 years old in the period January 1995 through December 2005, free of previous VTE and current use of oral contraceptives.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Absolute incidence of thromboembolic event